CLINICAL TRIAL: NCT03376425
Title: Application of Transthoracic Shear-wave Ultrasound Elastography in the Diagnosis of Pulmonary Lesions
Brief Title: Transthoracic Shear-wave Ultrasound Elastography
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201709073RINB
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Elasticity Imaging Techniques
Keywords: Chest ultrasound,Lung tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This study aims to provide the information of tissue elasticity in different etiologies of pulmonary lesions and to validate the predictive value of shear-wave elastography in differentiating benign pulmonary lesions from malignant lesions.

ELIGIBILITY:
1. Inclusion criteria: (1) Retrospective cohort from Jan 2016 to Dec 2017 (2) Patients with radiographic evidence of pulmonary tumors
2. Exclusion criteria: (1) age < 20 y/o (2) patients who can't hold their breath for 5 seconds

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chest ultrasonography in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-12-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Application of Transthoracic Shear-wave Ultrasound Elastography in the Diagnosis of Pulmonary Lesions | six months
  to provide the information of tissue elasticity in different etiologies of pulmonary lesions and to validate the predictive value of shear-wave elastography in differentiating benign pulmonary lesions from malignant lesions

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Kuo YW, Chen YL, Wu HD, Chien YC, Huang CK, Wang HC. Application of transthoracic shear-wave ultrasound elastography in lung lesions. Eur Respir J. 2021 Mar 25;57(3):2002347. doi: 10.1183/13993003.02347-2020. Print 2021 Mar. PMID 33033150